CLINICAL TRIAL: NCT00225992
Title: A Phase II Research Study of Arsenic Trioxide (Trisenox) in Patients With Myelodysplastic Syndrome (MDS)
Brief Title: Phase II Research Study of Arsenic Trioxide (Trisenox) in Patients With Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to lack of accrual.
Sponsor: Oncology Specialties, Alabama (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CCI-MDS-04
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Arsenic Trioxide

SUMMARY:
In this phase II study besides evaluating for safety, the primary efficacy parameter is to evaluate the incidence of patients who have had a response to Trisenox by evidence of increased blood counts (red, white, or platelets) and/or by decrease or transfusion dependency. The secondary efficacy parameter is the assessment of the tolerability of the new dosing schedule.

Arsenic trioxide will be administered intravenously over 1 to 2 hours with a loading dose of 0.30mg/kg for days 1-5 of the first week and then twice weekly for 27 weeks for a total of 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Myelodysplastic Syndrome by FAB. Can be made with cytogenetic analysis of Bone Marrow or Hematologist evaluation
* Patient must have had bone marrow biopsy and aspiration to confirm diagnosis within 60 days prior to treatment
* ECOG performance status of 0-2
* An EKG must be performed within 7 days prior to treatment to confirm QT interval <460msec.
* Serum creatinine less than or equal to 2.5 times the upper limit of normal.
* Serum bilirubin less than or equal to 2.5 times the upper limit of normal.
* Serum potassium greater than or equal to 4.0 mEq/dL and serum magnesium greater than or equal to 1.8 mg/dL. If these serum electrolytes are below the specified limits on the baseline laboratory tests, electrolytes should be administered to bring the serum concentrations to these levels before administering arsenic trioxide.
* Patients must be 18 years of age to participate in this study

Exclusion Criteria:

* Pregnant or nursing women, and men or women of childbearing potential who are unwilling to employ adequate contraception.
* Corrected QT interval of greater than or equal to 460msec in the presence of serum potassium and magnesium values within normal range.
* Significant CHF, coronary is ischemia or serious Arrhythmias including conduction delays.
* Peripheral neuropathy greater than or equal to 2.
* Evidence of active infection
* Concurrent treatment with maintenance therapy, cytotoxic chemotherapy, radiation, or investigational agents.
* Inability or unwillingness to comply with the treatment protocol, follow up, or research tests.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. Waples, MD, Principal Investigator — Oncology Specialties, PC
Locations (2):
- United States (2):
  - Comprehensive Cancer Institute, Decatur, Alabama
  - Comprehensive Cancer Institute, Huntsville, Alabama

REFERENCES:
- See also: Comprehensive Cancer Institute — http://www.ccihsv.com